CLINICAL TRIAL: NCT03061838
Title: Multicenter Double-blind Randomized Clinical Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Biosimilar Drug Ritumax® Compared to Original Drug MabThera® in Patients With Rheumatoid Arthritis
Brief Title: Safety, Tolerability, PK and PD of Biosimilar Drug Ritumax® Compared to Original Drug MabThera®
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biointegrator LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONCRA-RXM-02
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MabThera® (Active Comparator): 2 intravenous infusions on Week 0 and Week 2 (14-day interval).
  Interventions: Drug: MabThera®
- Ritumax® (Experimental): 2 intravenous infusions on Week 0 and Week 2 (14-day interval).
  Interventions: Drug: Ritumax®

INTERVENTIONS:
Drug: MabThera® — 1000 mg intravenously
  Other Names: Rituximab
  Arms: MabThera®
Drug: Ritumax® — 1000 mg intravenously
  Arms: Ritumax®

SUMMARY:
This is a multicenter, double-blind, randomized clinical study of safety, tolerability, pharmacokinetics and pharmacodynamics of biosimilar drug Ritumax® compared to original drug MabThera® in patients with rheumatoid arthritis, receiving stable doses of Methotrexate.

At Week -2, after signing the Patient Information Sheet and Informed Consent Form, patients with rheumatoid arthritis receiving stable doses of Methotrexate (10-25 mg per week orally or parenterally) will pass screening procedures.

Patients meeting all the inclusion/exclusion criteria will be invited to the investigational site for Visit 2 (Week 0) to be randomized into one of two treatment arms:

* Ritumax® 1000 mg х 2 intravenous infusions
* MabThera® 1000 mg х 2 intravenous infusions After being assigned to the treatment arm patients will receive a course of study treatment, including two i/v infusions at 14-day interval: at Week 0 and Week 2.

After that, patients will be followed up for the next 22 weeks. Safety, pharmacokinetic and pharmacodynamic parameters will be monitored at this visits.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent Form to participate in the study.
2. Men and women aged 18 years and older.
3. Patient diagnosed with rheumatoid arthritis of at least 6-month duration, determined according to classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) (ACR-EULAR 2010) or the American College of Rheumatology (ACR1987) (in case if the diagnosis of rheumatoid arthritis was determined till 2010).
4. Active phase of the disease confirmed due to the combination of the following parameters:

   * DAS28 > 3,2
   * 5 (of 28) of tender and 5 (of 28) of swollen joints
   * CRP level ≥1,5 mg/dL and/or ESR > 28 mm/h
   * positive test for rheumatoid factor and/or CCP antibodies
5. Patients with negative response to or intolerability to the DMARD therapy.
6. Current outpatient therapy of rheumatoid arthritis:

   * continuous therapy with Methotrexate for at least 12 weeks prior to screening
   * stable doses of Methotrexate (10-25 mg per week) within 4 weeks prior to screening
   * when currently under the corticosteroids therapy, the dose should be stable within the last 4 weeks prior to screening and be less than 10 mg of Prednisolone or its equivalent
   * when currently under the NSAID therapy, the dose should be stable within the last 4 weeks prior to screening

Exclusion Criteria:

The patient will be deemed ineligible for the study meeting any of the following criteria:

1. Other inflammatory arthropathies apart from rheumatoid arthritis (e.g. gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme desease) or other system autoimmune diseases (e.g. systemic lupus erythematosus, inflammatory bowel disease, pneumosclerosis or Felly's syndrome, sclerodermia, inflammatory myopathy, mixed collagenosis or other crossed syndrome). Patients with secondary Sjorgen's syndrome or secondary limited cutaneous vasculitis with a rheumatoid arthritis background may participate in the study.
2. Chronic heart failure Class III or IV in New York Heart Association (NYHA) classification and clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation).
3. Serious chronic pulmonary diseases (COPD, bronchial asthma); functional dyspnea of severity level III and higher (due to the Medical Science Research Council scale for dyspnea).
4. Signs of significant uncontrolled concomitant disease, e.g. renal, hepatic, gastrointestinal, endocrine system and nervous system disorders, which, according to the Investigator's opinion, could prevent the patient's participation in the study.
5. Any surgical procedure, including bone and joint surgeries, or synovectomy (including arthrodesis or endoprosthesis replacement), performed within 12 weeks prior to screening or planned to be performed within 24 weeks after (except for small surgical procedures, requiring a local anesthesia or no anesthesia).
6. Infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | within a 24-week period
  Comparative assessment of pharmacokinetic parameters of Ritumax® and MabThera
Peak Plasma Concentration (Cmax) | within a 24-week period
  Comparative assessment of pharmacokinetic parameters of Ritumax® and MabThera

SECONDARY OUTCOMES:
CD19+ B- lymphocytes | within a 24-week period
  Comparative assessment of pharmacodynamic parameters of Ritumax® and MabThera®
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | within a 24-week period
  The number of patients with treatment-related AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "Scientific Research Institution of Rheumatology" Russian Academy of Medical Sciences (FSBI "SRIR" RAMS), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No